CLINICAL TRIAL: NCT02239250
Title: Assessing the Health Impact of Advance Water Filters and Improved Cookstoves in Western Province, Rwanda: A Cluster-randomised Controlled Trial
Brief Title: Water Filters and Improved Cookstoves in Western Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: DelAgua (Other); Emory University (Other); Portland State University (Other); University of Colorado, Boulder (Other); Oregon Health and Science University (Other); Ministry of Health, Rwanda (Other Government); National University, Rwanda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCT01882777_2
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2015-02

CONDITIONS: Diarrhoeal Disease; Respiratory Infection; Pneumonia
Keywords: Child health; Pneumonia; Diarrhoea; Household air pollution; PM2.5; Stove intervention; Biomass fuel; Monitoring and evaluation; Water filter; Compliance; Thermotolerant coliforms; Rwanda
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia; Diarrhea; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water filter and cookstove (Experimental): All household that appear on Government approved lists as belonging to ubudehe 1 & 2 categories in the 72 sectors randomised as intervention sectors will be eligible to receive one free water filtering device and one free cookstove. All households will be given instructions of how to use the intervention.
  Interventions: Device: Water filter and cookstove
- Control (No Intervention): All household that appear on Government approved lists as belonging to ubudehe 1 & 2 categories in the 24 sectors randomised as control sectors will continue with their traditional cooking methods and drinking practices.

INTERVENTIONS:
Device: Water filter and cookstove — The Vestergaard Frandsen Lifestraw Family™ 2.1 is a point-of-use water treatment system.Water is poured through a 20 micron pre-filter into a 6L influent water tank.This water then filters through a 0.20 micron hollow-fiber ultrafiltration membrane into a 5.5L storage container.Water is then poured through a plastic tap, which prevents re-contamination.This system filters up to 18,000L of water.The system exceeds the WHO's "highly protective" standard for household water treatment technologies.The EcoZoom™ Spartan stove concentrates the combustion process while channeling airflow to completely burn the fuel provided.The stove has a ceramic combustion chamber within a steel housing, which is topped with a cast iron stove.The stove includes a rack for placing firewood and a pot skirt that improves the thermal efficiency.The cookstoves and filters will be delivered together at no cost to participating households.Households will receive instructions on how to operate these devices.
  Other Names: Vestergaard Frandsen Lifestraw Family™ 2.1; EcoZoom™ Spartan
  Arms: Water filter and cookstove

SUMMARY:
DelAgua Health Rwanda (Implementation) Ltd. together with Rwanda Ministry of Health (MoH) are delivering an intervention, consisting on the free distribution of one advance water filter and one improved cookstove to all household classified as ubudehe 1 and 2 according to government approved registers (poorest tertile), in Western Province. The aim of this intervention is to reduce the morbidity and mortality associated with diarrhoeal diseases and pneumonia in Rwanda.

The London School of Hygiene and Tropical Medicine (LSHTM) will be undertaking an independent evaluation of this large-scale intervention to assess its impact on health. The trial will evaluate whether the provision of improved cookstoves and advance water filters can reduce pneumonia and diarrhoea disease in children under 5 years of age.

A cluster randomized controlled trial (CRCT) with two arms of unequal size (3:1 ratio) will be use to answer this question. The 96 sectors in Western Province, Rwanda, will be randomised to either receive the intervention or the control. Each eligible household in intervention sectors will receive one EcoZoom™ Spartan and one Vestergaard Frandsen Lifestraw Family™ 2.1 water filter free of charge. Eligible households in control sectors will continue with their traditional cooking and drinking practices. Health data on children under 5 years of age will be collected from community health worker (CHW) and health facility records all across Western Province to evaluate the health impact of the intervention. The study will encompass 12 months of follow-up. After this time the control sectors will receive the intervention.

This independent evaluation will also include a nested village-level study within the larger sector-level study, with the aim to evaluate uptake, consistent use and acceptability of the intervention, as well as to assess the impact on environmental exposures and health outcomes. 174 villages (74 controls and 74 intervention) will be selected for participation. Household surveys will be used to collect data on intervention use and acceptability as well as on self-reported health data. Water samples will be collected and monitoring of exposure to Households Air Pollution (HAP) will be undertaken. Measurements of blood pressure, expirated Carbon monoxide (CO) and pulse CO-oximetry will be undertake in primary cooks and or children under 5 years of age. Additionally, as part of this nested study, two exploratory studies will also be conducted. One will be focused on assessing the potential of biomarkers as indicators of environmental exposures (mainly HAP and water quality) and health status, while the other exploratory sub-study will assess the reactivity of participants to the use of remotely reporting electronic sensors to measure target behaviours.

ELIGIBILITY:
Inclusion Criteria:

* For Sector-level study:
* All households shown on updated 2012 government registers to be members of ubudehe 1 and 2 in Western Province, Rwanda will be eligible to participate in the study.
* For nested village-level study:
* All villages from all sectors in Western province, according to official Government lists will be eligible for participation with the exception of those villages that were selected for participation in Phase 1.
* At the village-level, all households that are classified as ubudehe 1 & 2 according to updated 2012 government registers, are part of the village, are able to provide informed consent, and that have at least one child under 4 years of age at the time of enrollment will be eligible for participation. Presence of a child under 4 years of age will be assessed by checking dates of birth or recorded age in months in the CHW register of children <5 years (Igitabo Cy'Ibikorwa Byo Gukurikirana), which are maintained at the village by CHW (though occasionally these are transferred to health centers). If this data is missing will be assesses based on CHW's report. In those cases where a village has more than the required number of participating households (10 household), a random selection of 10 households will be drawn.
* For the assessment of personal exposure to HAP a stricter set of eligibility criteria will be applied. Households that comply with the following eligibility criteria will be eligible for the exposure to HAP sub-study.

  * Have a child 1.5-4 year old,
  * Have a child healthy enough to wear the monitoring equipment (as perceived by the mother),
  * Have a non-smoking primary cook,
  * Have a primary cook that is currently not pregnant (as far as she is aware of), and
  * Have a primary cook that is in a healthy state to wear the monitoring equipment
* The first two households identified from a randomised list will be invited to participate.
* For the biomarker sub-studies, both the primary cook and the child under 4 years of age from households undergoing HAP exposure assessment will be eligible for the inflammatory cytokine biomarker study. For the enteric seroconversion study, all children aged 6 to 12 months will be eligible for participation.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1582 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of IMCI defined pneumonia in children under 5 years of age in ubudehe 1 & 2 categories | 12 months
  All types of pneumonia (severe, non severe). This outcome measure will be assessed in the sector-level study.
Incidence of IMCI defined diarrhoea in children under 5 years of age in ubudehe 1 & 2 categories | 12 months
  All types of diarrhoea (including severe, persistent, dysentery). This outcome measure will be assessed in the sector-level study.

SECONDARY OUTCOMES:
All-cause mortality in children under 5 years of age in ubudehe 1 & categories | 12 months
  This outcome measure will be assessed in the sector-level study.
Incidence of maternal health outcomes among women un ubudehe 1 & 2 categories | 12 months
  Incidence of maternal health outcomes including low birth weight, premature birth, and still birth
Prevalence of self-reported diarrhoea in children under 5 years of age in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Prevalence of pneumonia in children under 5 years of age in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.

OTHER OUTCOMES:
Prevalence of IMCI defined pneumonia in children under 5 years of age in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Prevalence of IMCI defined diarrhoea in children under 5 years of age in ubudehe 1 &2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Prevalence of self-reported diarrhoea among primary cooks | 12 months
  This outcome measure will be assessed in the nested village-level study.
Prevalence of self-reported respiratory conditions among primary cooks in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Mena difference in blood pressure in primary cooks in ubudehe 1 and 2 categories | 12 months
  Mean difference of systolic and diastolic measured separately. This outcome measure will be assessed in the nested village-level study.
Mean difference in levels of expirated CO in children under 5 years of age and primary cooks in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Mean difference levels of Carboxyhaemoglobin in children under 5 years of age and primary cooks in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Percentage seroconversion against enteric pathogens in children 6-12 months of age at enrolment in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Mean difference in inflammatory cytokines in children under 5 years of age in unudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Median difference in 48-h personal exposure to PM2.5 in children under 5 years of age and primary cooks in ubudehe 1 & 2 categories | 12 months
  This outcome measure will be assessed in the nested village-level study.
Levels of faecal contamination in drinking water | 12 months
  This outcome measure will be assessed in the nested village-level study. Proportion of water samples samples free of faecal contamination.
Levels of consistent use of the intervention | 12 months
  This outcome measure will be assessed in the intervention group only of the nested village-level study.
  Percentage of households reporting the use of the stove as their primary stove in all follow-up visits. Percentage of households reporting their current drinking water was treated by the intervention filter in all follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clasen, JD MSc PhD, Principal Investigator — LSHTM & Emory University
Locations (1):
- Manna Energy Ltd., Kigali, Kigali, Rwanda

REFERENCES:
- [Derived] Kirby MA, Nagel CL, Rosa G, Zambrano LD, Musafiri S, Ngirabega JD, Thomas EA, Clasen T. Effects of a large-scale distribution of water filters and natural draft rocket-style cookstoves on diarrhea and acute respiratory infection: A cluster-randomized controlled trial in Western Province, Rwanda. PLoS Med. 2019 Jun 3;16(6):e1002812. doi: 10.1371/journal.pmed.1002812. eCollection 2019 Jun. PMID 31158266
- [Derived] Nagel CL, Kirby MA, Zambrano LD, Rosa G, Barstow CK, Thomas EA, Clasen TF. Study design of a cluster-randomized controlled trial to evaluate a large-scale distribution of cook stoves and water filters in Western Province, Rwanda. Contemp Clin Trials Commun. 2016 Aug 2;4:124-135. doi: 10.1016/j.conctc.2016.07.003. eCollection 2016 Dec 15. PMID 29736475